CLINICAL TRIAL: NCT01862354
Title: Comparative Analgesic Effect Between Continuous Wound Infusion and Transverse Abdominal Plan Block for Abdominoplasty Surgery
Brief Title: Analgesic Effect Between TAP Block and Continuous Wound Infusion in Abdominoplasty Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, J P Lecoq, MD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-00017214-14 2013/9; 2013-000172-14 (EudraCT Number)
Record Dates: First submitted 2013-05-02; First posted 2013-05-24 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Surgery of Abdominoplasty With Flank Liposuction
Keywords: Postoperative analgesia; Abdominoplasty; Continuous wound infusion; Transverse abdominal plan block; Local anesthetics : Ropivacaine; Regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group TAP block (Active Comparator): Patients in this group received a transverse abdominal plan block with local anesthetics and clonidine as postoperative analgesia.
  Interventions: Procedure: Transverse abdominal plan block
- Group : Continuous wound infusion (Active Comparator): Patients in this group received continuous wound infusion with local anesthetics and clonidine as postoperative analgesia.
  Interventions: Procedure: Continuous wound infusion

INTERVENTIONS:
Procedure: Transverse abdominal plan block — Transverse abdominal plan block was performed after induction of anaesthesia and before surgery. 3 mg/kg of Ropivacaine 5mg/ml (maximum 200 mg) plus 150 microg of Clonidine were injected at the good place. The was realised with the aid of ultrasound
  Other Names: Regional anesthesia : TAP block
  Arms: Group TAP block
Procedure: Continuous wound infusion — In this group, a multihole catheter was surgically inserted vertically before skin closure. The catheter was primed with Ropivacaine 2 mg/ml 10 ml plus clonidine 150 microg before the end of anaesthesia. Continuous wound infusion was started at a rate of 10 ml per hour of Ropivacaine 2 mg/ml during the first 9 hours after the surgery.
  Other Names: Regional anesthesia : Continuous wound infusion
  Arms: Group : Continuous wound infusion

SUMMARY:
The purpose of this randomized controlled study is to compare the postoperative analgesic effect of a continuous wound infusion of local anesthetics and a sole transverse abdominal plan (TAP) regional block in the surgery of Abdominoplasty Combined With Flank Liposuction. Local anesthetics products used are ropivacaine combined with clonidine. Similar amount of local anesthetics and clonidine are used.

DETAILED DESCRIPTION:
In a first group, patients receive, after induction of anaesthesia and before surgery, a TAP block (transverse abdominal plan block) with 3mg/kg Ropivacaine 0.5% (maximum 200 mg) and 150 microg Clonidine.

In a second group, before skin closure, a multiholes catheter was inserted beyond the skin. 20 mg Ropivacaine 0.2% added with 150 microg Clonidine was injected as bolus dose through this catheter followed by a continuous infusion of Ropivacaine 0.2% 10ml per hour during the following 9 hours (total dose of 200 mgr).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for abdominoplasty combined with flank liposuction

Exclusion Criteria:

* Allergy to local anesthetics or clonidine
* Coagulation disorders
* History of chronic pain
* Alcohol or drugs dependance
* Refusal of the patients

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pain score expressed on a visual analogue scale | at 0,2,4,6, 8 hours, and day 1 and day 2 postoperatively

SECONDARY OUTCOMES:
Piritramide consumption on Patient Controlled Analgesia (PCA) device | at 0,2,4,6, 8 hours, and day 1 and day 2 postoperatively
Scale of nausea | at 0,2,4,6, 8 hours, and day 1 and day 2 postoperatively
  Scale of nausea was defined as :
  0 = No nausea - 1 = weak nausea - 2 = Moderate nausea - 3 = Important nausea
Scale of sedation | at 0,2,4,6, 8 hours, and day 1 and day 2 postoperatively
  Scale of sedation was defined as :
  0 = Awake patient - 1 = Quiet and awake - 2 = Sleepy but arousable - 3 = Sleepy and not arousable
Scale of patient's satisfaction | at day 2 postoperatively
  Scale of satisfaction was defined as :
  1 = Very satisfied - 2 = Satisfied with no enthusiasm - 3 = Not satisfied
Number of patients with adverse events | daily during 48 hours postoperatively

OTHER OUTCOMES:
Total of peroperative propofol consumption (mg) | at the end of the anesthesia (average time around 180 minutes)
Total of peroperative remifentanil consumption (mg) | at the end of the anesthesia (average time around 180 minutes)
Volume of peroperative liquid infiltrated (ml) | at the end of the surgery (average time around 150 minutes)
Volume of peroperative liquid suctioned (ml) | at the end of the surgery (average time around 150 minutes)
Weight of skin resection (mg) | At the end of the surgery (average time around 150 minutes)
Volume of surgical drainage (ml) | at day 1 and day 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre H Lecoq, Md, PhD, Principal Investigator — University of Liege, University Hospital
Locations (1):
- University of Liege, University Hospital, Liège, Belgium